CLINICAL TRIAL: NCT06138743
Title: A Phase 1/2a Dose-Escalating Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ARO-DM1 in Subjects With Type 1 Myotonic Dystrophy Who Are ≥18 to ≤ 65 Years
Brief Title: Study of ARO-DM1 in Subjects With Type 1 Myotonic Dystrophy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARODM1-1001; 2024-513579-42 (EudraCT Number)
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Myotonic Dystrophy 1
MeSH Terms: conditions — Myotonic Dystrophy | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- ARO-DM1 Intravenous (IV) Infusion (Experimental): Single or multiple doses of ARO-DM1 by IV infusion
  Interventions: Drug: ARO-DM1 Intravenous (IV) Infusion
- Placebo by IV Infusion (Placebo Comparator): Single or multiple doses of placebo by IV infusion
  Interventions: Drug: Placebo Intravenous (IV) Infusion
- ARO-DM1 Subcutaneous SC Injection (Experimental): Single or multiple doses of ARO-DM1 by sc injection
  Interventions: Drug: ARO-DM1 subcutaneous (SC) injection
- Placebo by SC Injection (Placebo Comparator): Single or multiple doses of placebo by sc injection
  Interventions: Drug: Placebo Subcutaneous (SC) Injection

INTERVENTIONS:
Drug: ARO-DM1 Intravenous (IV) Infusion — ARO-DM1 by intravenous (IV) infusion
  Arms: ARO-DM1 Intravenous (IV) Infusion
Drug: Placebo Intravenous (IV) Infusion — 0.9% NaCl calculated volume to match active treatment by IV infusion
  Arms: Placebo by IV Infusion
Drug: ARO-DM1 subcutaneous (SC) injection — ARO-DM1 by subcutaneous (SC) injection(s)
  Arms: ARO-DM1 Subcutaneous SC Injection
Drug: Placebo Subcutaneous (SC) Injection — 0.9% NaCl calculated volume to match active treatment by SC injection(s)
  Arms: Placebo by SC Injection

SUMMARY:
This is a phase 1/2a double-blinded, placebo-controlled, dose-escalating study to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of single and multiple ascending doses of ARO-DM1 compared to placebo in male and female subjects with type 1 myotonic dystrophy (DM1). Participants who have provided written informed consent and met all protocol eligibility requirements will be randomized to receive single (Part 1) or multiple (Part 2) doses of ARO-DM1 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed diagnosis of DM1
* Clinician-assessed signs of DM1 including clinically apparent myotonia
* Onset of DM1 symptoms occurred after the age of 12 years
* Walk for at least 10 meters independently at Screening
* Subjects of childbearing potential must agree to use highly effective contraception in addition to a condom during the study and for at least 90 days following the end of study or last dose of study drug, whichever is later. Subjects must not donate sperm or eggs during the study and for at least 90 days following the end of study or last dose of study drug whichever is later.

Exclusion Criteria:

* Inadequately controlled diabetes
* Confirmed diagnosis of congenital DM1
* Uncontrolled hypertension
* History of tibialis anterior (TA) biopsy within 3 months of Day 1 or planning to undergo TA biopsies during the study period
* Clinically significant cardiac, liver or renal disease
* HIV infection (seropositive) at Screening
* Seropositive for hepatitis B (HBV) or hepatitis C (HCV) at screening
* Untreated or poorly controlled epilepsy
* Treatment with anti-myotonia medication within a period of 5 half-lives of the medication prior to Screening.
* Abnormal coagulation parameters at Screening including platelet count, international normalized ratio (INR), prothrombin time, and activated partial thromboplastin time (APTT)

Note: Additional inclusion/exclusion criteria may apply per protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment -Emergent Adverse Events (TEAEs) Over Time Through End of Study (EOS) | Single-dose phase (Part 1): Up to Day 90(EOS); multiple-dose phase (Part 2): Up to Day 180(EOS)

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ARO-DM1: Maximum Observed Plasma Concentration (Cmax) | Single-dose phase (Part 1): Up 24 hours post-dose; multiple-dose phase (Part 2): Through 24 hours post first and second dose
PK of ARO-DM1: Area Under the Plasma Concentration Versus Time Curve from Zero to 24 Hours (AUC0-24) | Single-dose phase (Part 1): Up 24 hours post-dose; multiple-dose phase (Part 2): Through 24 hours post first and second dose
PK of ARO-DM1: Area Under the Plasma Concentration Versus Time Curve from Zero to the Last Quantifiable Plasma Concentration (AUClast) | Single-dose phase (Part 1): Up 24 hours post-dose; multiple-dose phase (Part 2): Through 24 hours post first and second dose
PK of ARO-DM1: Area Under the Plasma Concentration Versus Time Curve from Zero to Infinity (AUCinf) | Single-dose phase (Part 1): Up 24 hours post-dose; multiple-dose phase (Part 2): Through 24 hours post first and second dose
Change from Baseline at Day 120 for Video Hand Opening Time (vHOT) | (Part 2): Baseline, Day 120
Change from Baseline Over Time for the Timed Up and Go Test (TUG) Assessment | (Part 2): Baseline through EOS (up to 180 days)
Change from Baseline Over Time for the 10-Meter Walk/Run Test (10MWT) Assessment | (Part 2): Baseline through EOS (up to 180 days)
Change from Baseline Over Time for the Hand-held Quantitative Dynamometry Assessment | (Part 2): Baseline through EOS (up to 180 days)
Change from Baseline Over Time for the Video Hand Opening Time (vHOT) Assessment | (Part 2): Baseline through EOS (up to 180 days)
Change from Baseline Over Time for the Myotonic Dystrophy Type 1 Activity and Participation Scale (DM1-Activ-C) Assessment | (Part 2): Baseline through EOS (up to 180 days)
Change from Baseline Over Time for the Myotonic Dystrophy Health Index (MDHI) Assessment | (Part 2): Baseline through EOS (up to 180 days)

CONTACTS AND LOCATIONS:
Locations (10):
- Australia (4):
  - Research Site, Liverpool, New South Wales
  - Research Site, Birtinya, Queensland
  - Research Site, Herston, Queensland
  - Research Site, Melbourne, Victoria
- Research Site, Christchurch, New Zealand
- Taiwan (2):
  - Research Site, Taichung
  - Research Site, Taipei
- Thailand (3):
  - Research Site, Bangkok, Bangkok
  - Research Site, Hat Yai, Changwat Songkhla
  - Research Site, Lampang

IPD SHARING:
Plan to Share IPD: No